CLINICAL TRIAL: NCT07136974
Title: Comparing the Efficacy of TQB2102 and TCbHP in Neoadjuvant Treatment for HER2-positive Early Breast Cancer: A Randomized Phase II Clinical Trial.
Brief Title: Efficacy of TQB2102 Versus TCbHP in Neoadjuvant Therapy for HER2-positive Early Breast Cancer.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-025
Record Dates: First submitted 2025-07-15; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; HER2 + Breast Cancer
Keywords: HER2 positive; neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2102 group (Experimental): TQB2102 is administered intravenously at 6 mg/kg every 3 weeks for 6 cycles.
  Interventions: Drug: TQB2102
- TCbHP (Active Comparator): Docetaxel + carboplatin + trastuzumab + pertuzumab (every 3 weeks)
  Interventions: Drug: Docetaxel + Carboplatin + Trastuzumab +Pertuzumab

INTERVENTIONS:
Drug: TQB2102 — TQB2102 is administered intravenously at 6 mg/kg every 3 weeks for 6 cycles.
  Arms: TQB2102 group
Drug: Docetaxel + Carboplatin + Trastuzumab +Pertuzumab — Docetaxel 75 mg/m2(day 1) , Carboplatin (AUC=6) (day 1), Trastuzumab (8mg/kg first dose, 6mg/kg sequential) and Pertuzumab (840mg first dose, 420mg/kg sequential) are administered intravenously every 3 weeks for 6 cycles.
  Arms: TCbHP

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of TQB2102 compared to TCbHP in the neoadjuvant treatment of HER2-positive breast cancer. Participants will randomly assigned, in a 1:1 ratio, to receive either TQB2102 or TCbHP for 6 cycles. Patients will undergo definitive surgery (breast conservation or mastectomy with sentinel lymph-node evaluation or axillary dissection) 3 to 6 weeks after the last cycle of the neoadjuvant phase. Primary endpoint is pathological complete response, defined as pathological stage ypT0/Tis ypN0 at the time of definitive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years,
2. ECOG performance status 0-1;
3. Clinical T2-T4, or T1c with axillary lymph node metastasis; Confirmed HER2-positive status (per 2018 ASCO/CAP HER2 Testing Guidelines, defined as IHC 3+ or FISH positive);
4. Clinically measurable lesion: Lesion measurable by ultrasound, mammography, or optional MRI within 1 month before randomization;
5. No chemotherapy contraindications based on organ and bone marrow function tests within 1 month prior to chemotherapy: Absolute neutrophil count (ANC) ≥1.5×10⁹/L, Hemoglobin ≥90 g/L, Platelet count ≥100×10⁹/L, Total bilirubin <1.5 × ULN (upper limit of normal), Creatinine <1.5 × ULN, AST/ALT <1.5 × ULN, Echocardiography: Left ventricular ejection fraction (LVEF) ≥50%;
6. For women of childbearing potential: Negative serum pregnancy test within 14 days before randomization;
7. Signed informed consent form.

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer;
2. Prior treatments received including chemotherapy, endocrine therapy, targeted therapy, or radiotherapy; History of other malignancies within 3 years or concurrent malignancies. Exceptions: Other malignancies treated with surgery alone achieving ≥5-year disease-free survival (DFS) . Cured cervical carcinoma in situ or non-melanoma skin cancer;
3. Major non-breast cancer-related surgical procedures within 4 weeks prior to enrollment, or incomplete recovery from such procedures;
4. Significant cardiac disease or conditions including but not limited to: History of heart failure or systolic dysfunction (LVEF <50%). Uncontrolled high-risk arrhythmias: Atrial tachycardia, resting heart rate >100 bpm, significant ventricular arrhythmias (e.g., ventricular tachycardia), or high-grade atrioventricular block (Mobitz II second-degree or third-degree AV block). Angina requiring anti-anginal medication. Clinically significant valvular heart disease. ECG evidence of transmural myocardial infarction. Poorly controlled hypertension (SBP >180 mmHg and/or DBP >100 mmHg);
5. Contraindications to chemotherapy per investigator's assessment due to severe uncontrolled comorbidities;
6. Known hypersensitivity to protocol drug components;
7. History of immunodeficiency disorders (including HIV positivity), other acquired/congenital immune deficiencies, or organ transplantation;
8. Any concurrent condition that in the investigator's judgment would jeopardize patient safety or compromise study completion, or other grounds for ineligibility.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-08-30 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | up to 180 days
  pCR was defined as ypT0/Tis ypN0 at surgery

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | 5-10 years
  EFS was defined as time from randomization to invasive progression (local/distant), recurrence, or death.
Adverse Event (AE) | up to 180 days
Overall Survival (OS) | 5-10 years
  OS was measured from randomization to death from any cause. Patients without documented death were censored at the last contact date.
Objective Response Rate （ORR） | up to 180 days

OTHER OUTCOMES:
PCR in Pre-Specified subgroup analysis | up to 180 days
  PCR in subgroups defined by HR status，HER2 IHC and clinical stages

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided